CLINICAL TRIAL: NCT00508378
Title: Chemotherapy-Related Toxicities In Ovarian Cancer Patients: Preference Assessments of Patients, Family Members, Ancillary Staff and Gynecologic Oncologists, and Patients' Quality of Life
Brief Title: Chemotherapy-Related Toxicities In Ovarian Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: GYN00-409
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Quality of Life; Chemotherapy Side-Effects; Interview; Questionnaire; Caregivers
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Interview & Questionnaires
  Interventions: Behavioral: Interview; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Interview — Interview regarding side-effects of chemotherapy, 30-45 minutes.
  Other Names: Survey
Behavioral: Questionnaire — Quality of life survey and symptom assessment questionnaire, 15 minutes.

SUMMARY:
Primary Objectives:

1. To assess the preferences of women with ovarian cancer, their clinical caregivers, familial caregivers, and a control group for toxicities associated with chemotherapy.

   * To compare preferences of women with ovarian cancer to preferences of their clinical caregivers.
   * To compare preferences of women with ovarian cancer to preferences of their familial caregivers.
   * To compare preferences of women with ovarian cancer to preferences of a women in the control group.
2. To prospectively collect quality of life data from women with ovarian cancer.
3. To prospectively collect symptom assessment data from women with ovarian cancer.

DETAILED DESCRIPTION:
Patients in this study will be recruited from the Gynecologic Oncology Clinic waiting area. All participants (patients, family and clinical caregivers, control group women with no cancer) in this study will take part in an interview to see how they feel about the different side-effects of chemotherapy. The interview will involve reading short descriptions of the side-effects and then answering some questions that ask for an opinion. The actual interview will take about 30-45 minutes to complete. The interviews will either take place in private conference rooms in the clinic or in private rooms at the Ambulatory Treatment Center (ATC).

Patients will also be given quality of life and symptom assessment questionnaires. The questionnaires are simple to read and quick to answer. The questionnaire takes about 15 minutes to complete.

The participant's involvement in this study is limited to the questionnaire/interview. Once that is done, the participant is finished with the study.

This is an investigational study. A total of 288 people will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Women with epithelial ovarian cancer presenting to the UTMDACC Gynecologic Oncology Clinic who are currently undergoing chemotherapy
2. Women with a history of epithelial ovarian cancer presenting to the UTMDACC Gynecologic Oncology Clinic who are seen in follow-up
3. Women who are at least 18 years of age
4. Women who speak English
5. Clinical caregivers of patients with ovarian cancer (UTMDACC gynecologic oncologists, UTMDACC gynecologic medical oncologists, UTMDACC registered nurses and licensed vocational nurses in the UTMDACC Gynecology Clinic, and UTMDACC gynecologic oncology fellows and residents)
6. Familial caregivers of patients with ovarian cancer (primary caregiver)

Exclusion Criteria:

1. Participants who are non-English speakers
2. Participants who are less than 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ovarian cancer patients, their family members, and doctors and nurses from the UTMDACC Gynecologic Oncology Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2001-01 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Qualitative information on how ovarian cancer patients, their family members, and doctors and nurses feel about the side-effects of chemotherapy. | 8 Years

SECONDARY OUTCOMES:
Patient Response to Quality of Life Using Interview + Questionnaire | 30 minute interviews + 15 minutes for questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Diane C. Bodurka, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org